CLINICAL TRIAL: NCT00522288
Title: Adolescent and Child Health Initiative to Encourage Vision Empowerment (ACHIEVE) Study
Brief Title: Effects of Contact Lens Wear on Children's Self-Perceptions
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Jeffrey J. Walline, OD, PhD, College of Optometry, The Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2003H0114
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Myopia
Keywords: Myopia; Self-Perception; Contact Lenses; Glasses; Randomized; Children; Self-esteem
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic; Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contact Lens (Experimental): Soft contact lenses
  Interventions: Device: Soft contact lenses
- Spectacle (Active Comparator): Spectacles
  Interventions: Device: Spectacle

INTERVENTIONS:
Device: Soft contact lenses — Daily wear soft contact lenses disposed of daily or biweekly
  Other Names: 1 Day Acuvue or Acuvue 2 contact lenses
  Arms: Contact Lens
Device: Spectacle — Spectacles for the treatment of myopia
  Other Names: Children chose their own frames.
  Arms: Spectacle

SUMMARY:
The purpose of the study is to determine whether contact lens wear will improve children's self-perceptions more than spectacle wear.

DETAILED DESCRIPTION:
Eight to eleven year old children will be randomly assigned to wear spectacles or soft contact lenses. The children's self-perceptions will be measured at baseline and every six months. We will compare the change in self-perception between spectacle and soft contact lens wearers over three years. We will also examine the effect of how much children initially like or dislike to wear glasses on the change in self-perception over three years.

ELIGIBILITY:
Inclusion Criteria:

* 1.00 to 6.00 D spherical component myopia, based on cycloplegic autorefraction
* 1.00 DC or less astigmatism, based on cycloplegic autorefraction
* 20/20 or better best-corrected visual acuity in each eye
* Global stereoacuity of 250 seconds of arc or better based on Randot stereoacuity

Exclusion Criteria:

* Contact lens wear within the past month
* Ocular health problems that could affect vision, eye development, or contact lens wear
* Systemic health problems that could affect understanding of surveys or contact lens wear
* Participation in other eye or vision studies that prescribed a treatment

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 484 (Actual)
Dates: Start 2003-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Global Self-Worth Scale from the Self-Perception Profile for Children | 3 years

SECONDARY OUTCOMES:
Five other scales from the Self-Perception Profile for Children | 3 years
Change in cycloplegic autorefraction | 3 years
Change in axial length, measured by A-scan ultrasound | 3 years
Change in corneal curvature, measured by Grand Seiko WR-5100K autokeratometer | 3 years
Change in Overall score from the Pediatric Refractive Error Profile | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Walline, OD, PhD, Principal Investigator — Ohio State University
Locations (5):
- United States (5):
  - New England College of Optometry, Boston, Massachusetts
  - Ohio State University College of Optometry, Columbus, Ohio
  - Pacific University College of Optometry, Forest Grove, Oregon
  - Southern College of Optometry, Memphis, Tennessee
  - University of Houston College of Optometry, Houston, Texas

REFERENCES:
- [Background] Walline JJ, Jones LA, Chitkara M, Coffey B, Jackson JM, Manny RE, Rah MJ, Prinstein MJ, Zadnik K. The Adolescent and Child Health Initiative to Encourage Vision Empowerment (ACHIEVE) study design and baseline data. Optom Vis Sci. 2006 Jan;83(1):37-45. doi: 10.1097/01.opx.0000195566.94572.eb. PMID 16432471
- [Background] Walline JJ, Long S, Zadnik K. Daily disposable contact lens wear in myopic children. Optom Vis Sci. 2004 Apr;81(4):255-9. doi: 10.1097/00006324-200404000-00011. PMID 15097767
- [Result] Walline JJ, Jones LA, Sinnott L, Chitkara M, Coffey B, Jackson JM, Manny RE, Rah MJ, Prinstein MJ; ACHIEVE Study Group. Randomized trial of the effect of contact lens wear on self-perception in children. Optom Vis Sci. 2009 Mar;86(3):222-32. doi: 10.1097/OPX.0b013e3181971985. PMID 19214129
- [Result] Walline JJ, Jones LA, Sinnott L, Manny RE, Gaume A, Rah MJ, Chitkara M, Lyons S; ACHIEVE Study Group. A randomized trial of the effect of soft contact lenses on myopia progression in children. Invest Ophthalmol Vis Sci. 2008 Nov;49(11):4702-6. doi: 10.1167/iovs.08-2067. Epub 2008 Jun 19. PMID 18566461
- [Result] Rah MJ, Walline JJ, Jones-Jordan LA, Sinnott LT, Jackson JM, Manny RE, Coffey B, Lyons S; ACHIEVE Study Group. Vision specific quality of life of pediatric contact lens wearers. Optom Vis Sci. 2010 Aug;87(8):560-6. doi: 10.1097/OPX.0b013e3181e6a1c8. PMID 20562669
- [Result] Jones-Jordan LA, Chitkara M, Coffey B, Jackson JM, Manny RE, Rah MJ, Walline JJ. A comparison of spectacle and contact lens wearing times in the ACHIEVE study. Clin Exp Optom. 2010 May;93(3):157-63. doi: 10.1111/j.1444-0938.2010.00480.x. PMID 20557557
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645